CLINICAL TRIAL: NCT00962416
Title: Comparison of Biolimus Eluted From an Erodable Stent Coating With Bare-Metal Stents in Acute ST-Elevation Myocardial Infarction and In Vivo 3-Vessel Assessment of Time-Related Changes of Culprit and Non-Culprit Lesions by IVUS/OCT in AMI
Brief Title: Comparison of Biomatrix Versus Gazelle in ST-Elevation Myocardial Infarction (STEMI)
Acronym: COMFORTABLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Prof. Stephan Windecker, Cardiology Department, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 137/09; 1373 (Other: Inselspital)
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Drug eluting stent; Biolimus; Biodegradable stent; ST-elevation myocardial infarction; Coronary artery disease
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Biolimus eluting Stent (Biomatrix)
  Interventions: Device: Biolimus eluted from an erodable stent coating (Biomatrix)
- 2 (Active Comparator): Bare metal stent (Gazelle)
  Interventions: Device: bare-metal stent (Gazelle)

INTERVENTIONS:
Device: Biolimus eluted from an erodable stent coating (Biomatrix) — The Biolimus-eluting stent (Biomatrix) has a corrugated ring design available in six and nine cell models and is laser cut from 316L VM stainless steel hypotube. The nominal dosage of Biolimus A9 goes from 133 to 442 microgram. The producer of the drug is Nippoon Kayaku Co., Ltd Takasaki Plant, 239, Iwahanamachi, Takasaki-shi, Gumma 370-1028 Japan. The biodegradable polymer is polylactic acid, which has become one of the most commonly used biodegradable polymers. Polylactic acid, its co-polymers, and mixtures have been evaluated in the preclinical, and clinical studies, revealing a favorable biocompatability profile. The polymer has been demonstrated to be safe when used as implant of drug release-control polymer for both animals and humans.
  Arms: 1
Device: bare-metal stent (Gazelle) — A bare-metal stent of identical design without surface application of polymer and drug.
  Arms: 2

SUMMARY:
Stent study:

Treatment of patients with acute myocardial infarction with drug eluting stents (DES) is effective but there remain concerns regarding the long-term safety and adverse effects on the adjacent arterial wall. The biolimus-eluting Biomatrix stent addresses the issues by incorporating modifications as a biodegradable polymer and a drug application solely to the abluminal stent surface. While clinical data about the biolimus-eluting stent show a favorable safety and efficacy profile, they require confirmation in a dedicated randomised trial in the subset of patients with STEMI. Therefore, the study is designed to compare the safety and efficacy of biolimus-eluting Biomatrix stent as compared to a bare metal stent of otherwise identical design in a prospective, multicenter, randomized, controlled superiority trial in patients with acute ST-elevation myocardial infarction.

Stent and Plaque Imaging Substudy:

In a substudy of the above mentioned stent trial, the investigators will perform a prospective, multicenter, longitudinal cohort study of 100 consecutive STEMI patients undergoing urgent coronary angiography and will employ high-resolution Optical Coherence Tomography (OCT) imaging technology and intra-vascular ultrasound and virtual histology (IVUS-VH) of the culprit STEMI lesions pre- and postprocedural as well as at a 13 months follow up. Assessment of vascular wall responses, including volumetric measurements of vessel, stent, lumen, peri-stent plaque, and intimal hyperplasia, indices of remodeling, stent expansion, and stent-vessel wall apposition in response to biolimus-eluting and bare-metal stent implantation will be performed. Moreover, IVUS, IVUS-VH and OCT will be performed in all three epicardial vessels in order to quantify and map the number, frequency and distribution of ruptured plaques at baseline and follow-up and quantify the morphological changes of ruptured and vulnerable plaques at baseline and follow-up and quantify the morphological changes over time in response to standard medical treatment. Therefore, new insight regarding the frequency, distribution, composition and evolution of coronary artery plaques and their prognostic impact on patients clinical outcome can be expected from the present study. Since patients suffer from a recurrent ischemic event rate of 5-10% during the first year, these findings may have important therapeutic implications for the medical treatment of affected patients to further reduce the risk of recurrence and improve prognosis.

DETAILED DESCRIPTION:
Background

Stent Study:

A routine invasive strategy using percutaneous coronary intervention (PCI) has been shown to improve survival and freedom from recurrent myocardial infarction compared to a thrombolysis in patients with acute ST-elevation myocardial infarction (STEMI). In addition to standard medical treatment, PCI with the use of coronary artery stents not only eliminate the underlying stenotic lesion, but afford a mechanical mean of plaque stabilization, normalize coronary blood flow, reduce shear stress, and local intracoronary thrombosis. Notwithstanding, the implantation of coronary artery stents is associated with arterial injury initiating a vasculo-proliferative cascade and as a result provoke structural changes of the vessel wall. The implantation of bare-metal stents (BMS) during primary percutaneous coronary interventions (P-PCI) in STEMI patients resulted in restenosis in up to 20% of patients and has not been shown to reduce the rate of mortality and reinfarction. Randomised trials and meta-analyses showed that the use of drug-eluting stents (DES) compared with BMS in patients with STEMI significantly reduces the rate of target lesion revascularization (TLR) without negative impact on the rate of death and myocardial infarction up to one year.

However, there remain important caveats surrounding the safety of DES in patients with STEMI and evidence of harm may only arise during longer term follow up. DES implantation into culprit lesions of patients with acute coronary syndromes has been identified as independent predictor of late stent thrombosis. DES as opposed to BMS implanted into a pro-thrombotic, inflammatory milieu of ruptured plaques in STEMI patients may lead to aneurysmal changes of the adjacent vessel wall. First generation DES implanted into STEMI lesions were found to be associated with substantial delay in healing compared to BMS. Moreover, DES implanted into STEMI lesions have been associated with a higher frequency of incompletely apposed struts and uncovered struts as assessed by OCT compared with DES implanted into stable lesions. These data suggest a significantly increased risk of late thrombotic complications related to DES. The phenomenon of aneurysmal change of the vessel wall may lead to incomplete stent apposition, which in turn may predispose to late complications such as stent thrombosis, recurrent myocardial infarction, and death. In conclusion, although coronary artery stents constitute a routine medical intervention to improve the acute and long-term result in STEMI patients, only very limited information exists as to the long-term clinical outcome and structural changes of the adjacent vessel wall.

First generation DES with controlled release of sirolimus or paclitaxel from durable polymers have reduced angiographic and clinical measures of restenosis in patients with STEMI. Limus analogues are more effective as site-specific agents than paclitaxel to reduce neointimal growth and repeat revascularisation procedures. However, late stent thrombosis is more germane to first-generation drug-eluting stents than to bare-metal stents owing to delayed healing and re-endothelialization. Furthermore, hypersensitivity reactions from the polymers may further increase the risk of stent thrombosis. These effects may be particularly pronounced in ruptured plaques of STEMI patients due to the direct contact with the necrotic core.

The biolimus-eluting stent to be studied in the present proposal has several features, which attenuate the above mentioned adverse effects. First, the polymer-drug combination is applied solely to the abluminal stent strut surface (rather than circumferential), thus maximizing the exposure to the vessel wall while minimizing release into the circulation. Second, the drug (biolimus A9) is released from a biodegradable polymer, which completely degrades into carbondioxide and water during a 6-9 months period, rendering the stent more closely to a BMS. Recently, the safety and efficacy of the biolimus-eluting stent using a biodegradable polymer was demonstrated in a large trial of 1,707 patients undergoing PCI. While the overall results showed non-inferiority for all safety and efficacy endpoints as compared with the sirolimus-eluting stent, the biolimus-eluting stent showed improved outcome in terms of MACE, stent thrombosis and TLR in the pre-specified subgroup of STEMI patients.

While clinical data as described above show a favorable safety and efficacy profile, the promising results ot the subgroup analysis require confirmation in a dedicated randomized trial in the subset of patients with STEMI. The present study is therefore designed to compare the safety and efficacy of the biolimus-eluting Biomatrix stent with a bare-metal stent of otherwise identical design in a prospective, multi-center, randomized, controlled trial in patients with acute ST-elevation myocardial infarction. To address the issue of late acquired stent apposition and stent strut coverage, an imaging substudy using grayscale IVUS and OCT will be performed.

Imaging Substudy:

A) Stent Imaging Substudy The implantation of drug eluting stents into a pro-thrombotic, inflammatory milieu of ruptured plaque in STEMI patients may lead to aneurysmal changes of the adjacent vessel wall possibly leading to incomplete stent apposition, which in turn may constitute a risk factor for late complications with adverse outcome. Delayed and incomplete stent strut coverage and endothelialization is another vessel wall reaction and possibly related to adverse late outcome by increasing the risk of late stent thrombosis. OCT provides a valuable modality for the assessment of stent strut coverage with 10x higher resolution than IVUS. Recently, biolimus-eluting stents have been shown to result in more complete stent strut coverage after 9 months as compared to sirolimus-eluting stents in the OCT substudy of the LEADERS trial. To compare the biological behaviour of a newer generation DES with biodegradable polymer as compared to a bare-metal stent, an imaging substudy using IVUS and OCT for detailed analyses of the post-procedural and follow-up vessel wall behaviour will be performed.

B)Plaque Imaging Substudy Although the short-term outcome of patients with ACS and STEMI has improved in recent years, clinical outcome at one year remains complicated by recurrent myocardial infarction and death in 10-15% of patients. Previous studies using angioscopy suggest delayed plaque healing, persistent thrombus, and recurrent plaque rupture as principal mechanisms for lesion progression and its clinical complications. However, these studies are limited by a small sample size, omission of follow-up imaging, lack of correlation with easily accessible serum markers, and unavailability of high resolution imaging technology such as OCT. Moreover, it is estimated that patients with ACS have more than one ruptured plaque in >40-80% of cases, which frequently are left untreated and therefore may contribute to long-term adverse clinical outcome.

Frequency, distribution, composition (TCFA versus non TCFA), and time-related changes of plaques of the entire coronary tree in patients with STEMI have not been documented so far, mainly due to technical limitations of the OCT imaging method. New-generation OCT systems available for the present study will allow the systematic assessment of long coronary segments. The combination of IVUS-VH and OCT will substantially improve the accuracy for detection of plaques and especially of TCFA.

Therefore, new insights regarding the frequency, distribution, composition and evolution of coronary artery plaques and their prognostic impact on patients clinical outcome can be expected from the present study. Since patients with ST-segment elevation myocardial infarction suffer from a recurrent ischemic event rate of 5-10% during the first year, these findings may have important therapeutic implications for the medical treatment of affected patients to further reduce the risk of recurrence and improve prognosis.

Objective

To establish superiority of the biolimus-eluting (Biomatrix) stent compared with an otherwise identical bare-metal stent (Gazelle) in terms of the composite endpoint of death, target-vessel related myocardial infarction at 1 year.

Imaging Substudy To compare neointimal thickness and strut coverage between both stent types in lesions of STEMI patients at 13 months and assessment of frequency, distribution and time related changes of culprit versus non culprit lesions of patients with acute ST-segment elevation myocardial infarction.

Methods

Stent study

This is a prospective, multi-center, randomized, assessor-blind, trial to be conducted at several swiss and european interventional cardiology sites. A total of 1100 patients will be randomized on a 1:1 basis to either the biolimus-eluting stent with biodegradable polymer or a bare-metal stent. The number of stents is not limited per patient, but it must be consistently implanted according to the assigned treatment allocation. All patients will be followed clinically for up to 5 years after stent implantation.

Imaging substudy

100 of 1100 randomized patients fulfilling the specific inclusion criteria (see above) will undergo IVUS-VH and OCT of the culprit lesions prior to and after stent implantation as well as during follow up. Moreover, IVUS-VH/OCT will be performed in all three major epicardial vessels at baseline and follow up. The imaging study will be performed at the University Hospital Bern, Geneva, Lausanne and Cardiocentro Lugano, all Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or more than 18 years
* Chest pain > 10 minutes
* Primary pci
* ST-segment elevation of > 1 mm in > 2 contiguous leads, or (presumably new) left bundle branch block, or true posterior MI with ST depression of > 1 mm in > 2 contiguous anterior leads
* Presence of at least one acute infarct artery target vessel with one or more coronary artery stenoses in a native coronary artery from 2.25-4 mm in diameter that can be covered with 1-multiple stents

Exclusion Criteria:

* Female of childbearing potential (age 50 and last menstruation within the last 12 months), who did not underwent tubal ligation, ovariectomy or hysterectomy
* Known intolerance to aspirin, clopidogrel, heparin, stainless steel, biolimus or contrast material
* Inability to provide informed consent
* Currently participating in another trial before reaching first endpoint
* Mechanical complication of acute myocardial infarction
* Acute myocardial infarction secondary to stent thrombosis
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the perisurgical period
* Noncardiac comorbid conditions are present with life expectancy 1 year or that may result in protocol malcompliance
* History of bleeding diathesis or known coagulopathy
* Use of Coumadin
* Additional for Imaging Substudy:

  * Age > 90 years
  * Hemodynamic instability
  * Renal failure
  * OCT/IVUS technically not feasible
  * Any patient in whom angiography demonstrates the infarct lesion to be at the site of a previously implanted stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1161 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACEs) in the overall population, defined as the composite of cardiac death, target-vessel related myocardial infarction (Q-wave and non-Q-wave), or ischemia-driven target lesion revascularization within 12 months | 30 days, 6 months, 1,2 and 5 years

SECONDARY OUTCOMES:
All deaths | 30 days, 6 months, 1,2 and 5 years
Clinically and non-clinically indicated target lesion revascularizations | 30 days, 6 months, 1, 2 and 5 years
Stent thrombosis ARC defined | 30 days, 1,2 and 5 years
Stent strut coverage as assessed by OCT | 13 months
Malapposition as assessed by OCT/IVUS | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, Professor of Cardiology, Study Chair — Dep. of Cardiology, University Hospital Bern; Lorenz Räber, MD, Study Director — Dep. of Cardiology, University Hospital Bern; Peter Jüni, Professor of Biostatistics, Study Director — Dep. of Social and Preventive Med., University Bern; Hector Garcia Garcia, MD, Study Director — Erasmus Thoraxcenter Rotterdam, The Netherlands
Locations (5):
- Switzerland (5):
  - Department of Cardiology, Bern
  - Dep. of Cardiology, Geneva
  - Dep. of Cardiology, Lugano
  - Dep. of Cardiology, University of Lausanne
  - Dep. of Cardiology, Zurich

REFERENCES:
- [Background] Costa RA, Lansky AJ, Abizaid A, Mueller R, Tsuchiya Y, Mori K, Cristea E, Leon MB, Sousa JE, Schmidt T, Hauptmann KE, Grube E. Angiographic results of the first human experience with the Biolimus A9 drug-eluting stent for de novo coronary lesions. Am J Cardiol. 2006 Aug 15;98(4):443-6. doi: 10.1016/j.amjcard.2006.02.051. Epub 2006 Jun 23. PMID 16893694
- [Background] Stone GW, Lansky AJ, Pocock SJ, Gersh BJ, Dangas G, Wong SC, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Mockel M, Ochala A, Kellock A, Parise H, Mehran R; HORIZONS-AMI Trial Investigators. Paclitaxel-eluting stents versus bare-metal stents in acute myocardial infarction. N Engl J Med. 2009 May 7;360(19):1946-59. doi: 10.1056/NEJMoa0810116. PMID 19420364
- [Result] Windecker S, Serruys PW, Wandel S, Buszman P, Trznadel S, Linke A, Lenk K, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Davies S, van Geuns RJ, Eerdmans P, van Es GA, Meier B, Juni P. Biolimus-eluting stent with biodegradable polymer versus sirolimus-eluting stent with durable polymer for coronary revascularisation (LEADERS): a randomised non-inferiority trial. Lancet. 2008 Sep 27;372(9644):1163-73. doi: 10.1016/S0140-6736(08)61244-1. Epub 2008 Aug 31. PMID 18765162
- [Derived] Bass RD, Garcia-Garcia HM, Ueki Y, Holmvang L, Pedrazzini G, Roffi M, Koskinas KC, Shibutani H, Losdat S, Ziemer PGP, Blanco PJ, Levine MB, Bourantas CV, Raber L. Effect of High-Intensity Statin Therapy on Atherosclerosis (IBIS-4): Manual Versus Automated Methods of IVUS Analysis. Cardiovasc Revasc Med. 2023 Sep;54:33-38. doi: 10.1016/j.carrev.2023.04.007. Epub 2023 Apr 15. PMID 37087308
- [Derived] Ueki Y, Yamaji K, Losdat S, Karagiannis A, Taniwaki M, Roffi M, Otsuka T, Koskinas KC, Holmvang L, Maldonado R, Pedrazzini G, Radu MD, Dijkstra J, Windecker S, Garcia-Garcia HM, Raber L. Discordance in the diagnostic assessment of vulnerable plaques between radiofrequency intravascular ultrasound versus optical coherence tomography among patients with acute myocardial infarction: insights from the IBIS-4 study. Int J Cardiovasc Imaging. 2021 Oct;37(10):2839-2847. doi: 10.1007/s10554-021-02272-6. Epub 2021 Jul 8. PMID 34236570
- [Derived] Bourantas CV, Raber L, Sakellarios A, Ueki Y, Zanchin T, Koskinas KC, Yamaji K, Taniwaki M, Heg D, Radu MD, Papafaklis MI, Kalatzis F, Naka KK, Fotiadis DI, Mathur A, Serruys PW, Michalis LK, Garcia-Garcia HM, Karagiannis A, Windecker S. Utility of Multimodality Intravascular Imaging and the Local Hemodynamic Forces to Predict Atherosclerotic Disease Progression. JACC Cardiovasc Imaging. 2020 Apr;13(4):1021-1032. doi: 10.1016/j.jcmg.2019.02.026. Epub 2019 Jun 12. PMID 31202749
- [Derived] Bourantas CV, Zanchin T, Sakellarios A, Karagiannis A, Ramasamy A, Yamaji K, Taniwaki M, Heg D, Moschovitis A, Fotiadis D, Mihalis L, Baumbach A, Torii R, Serruys P, Garcia-Garcia HM, Windecker S, Raber L. Implications of the local haemodynamic forces on the phenotype of coronary plaques. Heart. 2019 Jul;105(14):1078-1086. doi: 10.1136/heartjnl-2018-314086. Epub 2019 Mar 15. PMID 30877239
- [Derived] Raber L, Yamaji K, Kelbaek H, Engstrom T, Baumbach A, Roffi M, von Birgelen C, Taniwaki M, Moschovitis A, Zaugg S, Ostojic M, Pedrazzini G, Karagiannis-Voules DA, Luscher TF, Kornowski R, Tuller D, Vukcevic V, Heg D, Windecker S. Five-year clinical outcomes and intracoronary imaging findings of the COMFORTABLE AMI trial: randomized comparison of biodegradable polymer-based biolimus-eluting stents with bare-metal stents in patients with acute ST-segment elevation myocardial infarction. Eur Heart J. 2019 Jun 21;40(24):1909-1919. doi: 10.1093/eurheartj/ehz074. PMID 30851032
- [Derived] Koskinas KC, Zanchin T, Klingenberg R, Gencer B, Temperli F, Baumbach A, Roffi M, Moschovitis A, Muller O, Tuller D, Stortecky S, Mach F, Luscher TF, Matter CM, Pilgrim T, Heg D, Windecker S, Raber L. Incidence, Predictors, and Clinical Impact of Early Prasugrel Cessation in Patients With ST-Elevation Myocardial Infarction. J Am Heart Assoc. 2018 Apr 13;7(8):e008085. doi: 10.1161/JAHA.117.008085. PMID 29654204
- [Derived] Raber L, Klingenberg R, Heg D, Kelbaek H, Roffi M, Tuller D, Baumbach A, Zanchin T, Carballo D, Ostojic M, Stefanini GG, Rodondi N, von Birgelen C, Moschovitis A, Engstrom T, Gencer B, Auer R, Meier B, Mach F, Luscher TF, Juni P, Matter CM, Windecker S; COMFORTABLE and SPUM-ACS Trial Investigators. Safety of Prasugrel Loading Doses in Patients Pre-Loaded With Clopidogrel in the Setting of Primary Percutaneous Coronary Intervention: Results of a Nonrandomized Observational Study. JACC Cardiovasc Interv. 2015 Jul;8(8):1064-1074. doi: 10.1016/j.jcin.2015.03.023. PMID 26205445
- [Derived] Klingenberg R, Heg D, Raber L, Carballo D, Nanchen D, Gencer B, Auer R, Jaguszewski M, Stahli BE, Jakob P, Templin C, Stefanini GG, Meier B, Vogt P, Roffi M, Maier W, Landmesser U, Rodondi N, Mach F, Windecker S, Juni P, Luscher TF, Matter CM. Safety profile of prasugrel and clopidogrel in patients with acute coronary syndromes in Switzerland. Heart. 2015 Jun;101(11):854-63. doi: 10.1136/heartjnl-2014-306925. Epub 2015 Mar 20. PMID 25794517
- [Derived] Taniwaki M, Radu MD, Garcia-Garcia HM, Heg D, Kelbaek H, Holmvang L, Moschovitis A, Noble S, Pedrazzini G, Saunamaki K, Dijkstra J, Landmesser U, Wenaweser P, Meier B, Stefanini GG, Roffi M, Luscher TF, Windecker S, Raber L. Long-term safety and feasibility of three-vessel multimodality intravascular imaging in patients with ST-elevation myocardial infarction: the IBIS-4 (integrated biomarker and imaging study) substudy. Int J Cardiovasc Imaging. 2015 Jun;31(5):915-26. doi: 10.1007/s10554-015-0631-0. Epub 2015 Feb 28. PMID 25721728
- [Derived] Raber L, Taniwaki M, Zaugg S, Kelbaek H, Roffi M, Holmvang L, Noble S, Pedrazzini G, Moschovitis A, Luscher TF, Matter CM, Serruys PW, Juni P, Garcia-Garcia HM, Windecker S; IBIS 4 (Integrated Biomarkers and Imaging Study-4) Trial Investigators (NCT00962416). Effect of high-intensity statin therapy on atherosclerosis in non-infarct-related coronary arteries (IBIS-4): a serial intravascular ultrasonography study. Eur Heart J. 2015 Feb 21;36(8):490-500. doi: 10.1093/eurheartj/ehu373. Epub 2014 Sep 2. PMID 25182248
- [Derived] Taniwaki M, Stefanini GG, Raber L, Brugaletta S, Cequier A, Heg D, Iniguez A, Kelbaek H, Serra A, Ostoijic M, Hernandez-Antolin R, Baumbach A, Blochlinger S, Juni P, Mainar V, Sabate M, Windecker S. Predictors of adverse events among patients undergoing primary percutaneous coronary intervention: insights from a pooled analysis of the COMFORTABLE AMI and EXAMINATION trials. EuroIntervention. 2015 Aug;11(4):391-8. doi: 10.4244/EIJY14M07_12. PMID 25042419
- [Derived] Raber L, Kelbaek H, Ostojic M, Baumbach A, Heg D, Tuller D, von Birgelen C, Roffi M, Moschovitis A, Khattab AA, Wenaweser P, Bonvini R, Pedrazzini G, Kornowski R, Weber K, Trelle S, Luscher TF, Taniwaki M, Matter CM, Meier B, Juni P, Windecker S; COMFORTABLE AMI Trial Investigators. Effect of biolimus-eluting stents with biodegradable polymer vs bare-metal stents on cardiovascular events among patients with acute myocardial infarction: the COMFORTABLE AMI randomized trial. JAMA. 2012 Aug 22;308(8):777-87. doi: 10.1001/jama.2012.10065. PMID 22910755
- [Derived] Raber L, Heo JH, Radu MD, Garcia-Garcia HM, Stefanini GG, Moschovitis A, Dijkstra J, Kelbaek H, Windecker S, Serruys PW. Offline fusion of co-registered intravascular ultrasound and frequency domain optical coherence tomography images for the analysis of human atherosclerotic plaques. EuroIntervention. 2012 May 15;8(1):98-108. doi: 10.4244/EIJV8I1A16. PMID 22580254
- [Derived] Raber L, Kelbaek H, Ostoijc M, Baumbach A, Tuller D, von Birgelen C, Roffi M, Pedrazzini G, Kornowski R, Weber K, Heg D, Matter C, Luscher T, Taniwaki M, Meier B, Juni P, Windecker S. Comparison of biolimus eluted from an erodible stent coating with bare metal stents in acute ST-elevation myocardial infarction (COMFORTABLE AMI trial): rationale and design. EuroIntervention. 2012 Apr;7(12):1435-43. doi: 10.4244/EIJV7I12A224. PMID 22301368